CLINICAL TRIAL: NCT05745298
Title: The Use of Functional Electrical Stimulation in Conjunction With Respiratory Muscle Training to Improve Unaided Cough in Individuals With Acute Spinal Cord Injury
Acronym: AFES and RMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Stephane Philippe-ratway, Speech Pathologist, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221081
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Acute Spinal Cord Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AFES and RMT Paraplegia Group (Experimental): Patients with a diagnosis of paraplegia will receive co-treatment with abdominal functional electrical stimulation (AFES) and respiratory muscle training (RMT) for 2 weeks.
  Interventions: Device: Xcite Clinical Station
- AFES and RMT Tetraplegia Group (Experimental): Patients with a diagnosis of tetraplegia will receive co-treatment with abdominal functional electrical stimulation (AFES) and respiratory muscle training (RMT) for 4 weeks.
  Interventions: Device: Xcite Clinical Station

INTERVENTIONS:
Device: Xcite Clinical Station — The abdominal functional electrical stimulation (AFES) will be conducted using the Xcite system. This is a battery-powered stimulator with up to 12 channels of cyclical stimulation. It is a task-specific modality to enhance mass practice during neurological re-education. The electrical stimulation will be applied to the abdominal and back muscles. In addition, participants will receive two specific respiratory muscle training exercises performed 3 days per week.

SUMMARY:
The overall objective of this study is to improve unaided cough with abdominal and latissimus dorsi functional electrical stimulation in conjunction with respiratory muscle training in individuals with acute spinal cord injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic and atraumatic C2- T12 Spinal cord injury (AIS A, B, and C motor incomplete and complete injuries) currently admitted to inpatient rehabilitation with an injury date < 12 months prior to enrollment
2. Positive response to electrical stimulation through a palpable contraction
3. Fluent in written and spoken English

Exclusion Criteria:

1. Individuals who do not meet inclusion criteria
2. Prisoners
3. Concurrent traumatic brain injury determined by Rancho level of cognitive functioning < VI
4. Individuals with open tracheostomy
5. Persons with pacemakers
6. Pregnant women
7. Persons with epilepsy
8. Open wounds or metal implants at site of electrode placement
9. Unresponsive to functional electrical stimulation
10. Current diagnosis or history of thoraco-abdomino-pelvic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2027-07-21 (Estimated); Study Completion 2027-09-21 (Estimated)

PRIMARY OUTCOMES:
Percentage change in peak cough flow (PCF) | one week pre-intervention and up to 4 weeks post-intervention
  Assessing the percentage change in peak cough flow as assessed by peak expiratory flow meter with a pillow face mask.
Percentage change in peak expiratory flow | one week pre-intervention and up to 4 weeks post-intervention
  Assessing the percentage change in peak expiratory flow as assessed by peak expiratory flow meter with a pillow face mask.

SECONDARY OUTCOMES:
Percentage change in forced expiratory volume in 1 second (FEV1) | one week pre-intervention and up to 4 weeks post-intervention
  Assessing the percentage change in forced expiratory volume in 1 second (FEV1) as measured by the spirobank II. Measured in Liters/minute.
Percentage change in forced vital capacity (FVC) | one week pre-intervention and up to 4 weeks post-intervention
  Assessing the percentage change in forced vital capacity (FVC) as measured by the spirobank II. Measured in Liters/minute.
Percentage change in maximum inspiratory pressure (MIP) | one week pre-intervention and up to 4 weeks post-intervention
  Assessing the percentage change in maximum inspiratory pressure (MIP) as measured by the MicroSpiro. Measured in Liters/minute.
Percentage change in maximum expiratory pressure (MEP) | one week pre-intervention and up to 4 weeks post-intervention
  Assessing the percentage change in maximum expiratory pressure (MEP) as measured by the MicroSpiro. Measured in Liters/minute.
Change in cough effectiveness as measured by Likert Scale | one week pre-intervention and up to 4 weeks post-intervention
  The 5-point Likert scale will be used to obtain a self-rated perception of cough effectiveness. The participant will be asked to rate how strong and how well secretions were cleared after coughing. The rating scale will range from 1=very poor; 2=poor; 3=fair, 4=good; 5= very good. A score of 4 or 5 is classified as effectively clearing secretions after coughing.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Philippe-Ratway, MS, CCC-SLP, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No